CLINICAL TRIAL: NCT07034677
Title: Treatment With Indapamide in Patients With Post-Surgical Hypoparathyroidism
Acronym: HYPOCARE treat
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lars Rejnmark (Other)
Responsible Party: Sponsor-Investigator, Lars Rejnmark, MD, Ph.D., DMSc, prof, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CTIS 2024-516000-41-01; 2024-516000-41-01 (EU CTIS Number)
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hypoparathyroidism Post-surgical
Keywords: hypoparathyroidism; indapamide; hypercalciuria
MeSH Terms: conditions — Hypoparathyroidism; Hypercalciuria | interventions — Indapamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indapamide (Active Comparator): 14 days with active drug Indapamide 1.5 mg/day
  Interventions: Drug: Indapamide 1.5 MG SR
- Placebo (Placebo Comparator): 14 days with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indapamide 1.5 MG SR — 14 days treatment with indapamide 1.5 mg/day compared to placebo
  Arms: Indapamide
Drug: Placebo — 14 days treatment with placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effect of daily treatment with Indapamide for 14 days on urinary calcium excretion in patients with post surgical hypoparathyroidisme.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of daily treatment with Indapamide for 14 days on urinary calcium excretion in patients with post surgical hypoparathyroidisme.

Patients will do weekly blood sampling and 24 hour urine collection every second week.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic post surgical hypoparathyroidism diagnosed > 1 year ago
2. Age ≥ 18 years
3. Require treatment with active vitamin D ≥ 1 µg/day
4. Ionized plasma calcium between 1.15-1.25 mmol/L
5. 25(OH)D vitamin ≥ 50 nmol/L
6. Plasma magnesium > 0.65 mmol/L
7. Able to read and understand Danish
8. Willing and able to sign the informed consent form

Exclusion Criteria:

1. Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m3
2. Active cancer or former (except thyroid and basal cell skin) cancer treatment < 1 year ago
3. Pregnancy, pregnancy plans, or breastfeeding < 1 year ago
4. Abnormal arterial pressure at time of screening defined as symptomatic hypotension or systolic blood pressure < 100 mmHg
5. Plasma potassium < 3.5 mmol/L
6. Any current disease that might affect the calcium metabolism such as but not limited to:

   1. Recent prolonged immobility
   2. Untreated diabetes (HbA1c > 53 mmol/mol)
   3. Severe liver disease or hepatic encephalopathy
   4. Untreated thyroid disease
7. Current disease that might affect gastrointestinal absorption
8. Use of medications such as lithium or diuretics within 4 weeks prior to start of treatment
9. Known allergy or sensitivity to Indapamide, its excipients or sulfonamides
10. Known galactosemia, lactase deficiency, or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Urinary calcium excretion | Day 15
  investigate the effect of daily treatment with Indapamide for 14 days compared to placebo on urinary calcium excretion in patients with chronic post-surgical hypoparathyroidism

SECONDARY OUTCOMES:
Ionized calcium | Day 15
  To assess if treatment with Indapamide can affect the level of ionized calcium in the blood during treatment with Indapamide and hereby reduce the need for supplementation with oral calcium and active vitamin D.
Sodium diet | Day 15
  assess the efficacy of a low sodium diet in the placebo period on plasma ionized calcium and on the 24-hour urinary calcium excretion in patients with hypoparathyroidism
Safety (blood pressure) | Day 15
  To assess the safety (blood pressure) of daily treatment with Indapamide for 14 days compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, CSR
Time Frame: start data is time of publication and end 5 years after publication
Access Criteria: By contacting the leading author of the publication in order to make a data sharing agreement, which should be signed. Proposal for agreement must contain planned analyses. Statistical analyses have to be approved by independent review before published. Data sharing agreement needs to be approved by the Technology Transfer Office (TTO), Aarhus University Hospital, Denmark